CLINICAL TRIAL: NCT04199871
Title: Improving Control of Alignment in Intermittent Exotropia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Principal Investigator, Eileen Birch, Senior Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2019-1430
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): dichoptic 3D movies
  Interventions: Other: dichoptic 3D movies
- Group 2 (Sham Comparator): dichoptic standard movies
  Interventions: Other: dichoptic 3D movies

INTERVENTIONS:
Other: dichoptic 3D movies — dichoptic movies presented on a Nintendo 3DS
  Other Names: dichoptic standard movies

SUMMARY:
Aim 1: To determine whether use of dichoptic movies for 4 weeks may be helpful in improving control of alignment in children with intermittent exotropia (IXT), thus allowing IXT to be managed non-surgically Aim 2: To determine pre-IXT surgery use of dichoptic movies for 4 weeks post-operatively may be helpful in maintaining successful control of alignment in children who have surgical correction of IXT

DETAILED DESCRIPTION:
The most common childhood-onset exotropia is intermittent exotropia (IXT). IXT is an exotropia that is not constant and is mainly present at distance, but may also be present at near. Binocular single vision is typically present at near but may be subnormal. There is some debate in the literature about whether or not these children should be treated surgically to correct the misalignment. It can be argued that prompt surgical correction is necessary to prevent the development of suppression of the deviating eye, progression to constant exotropia, and permanent changes in sensory function that may compromise long-term post-operative outcomes. On the other hand, statistics on the natural history of IXT suggest that progression to constant XT occurs in less than 25% and up to 15% may improve spontaneously. These findings suggest a more conservative approach, using surgery only if deterioration of the IXT occurs. A recent randomized clinical trial of the two most common surgical techniques for IXT revealed a 3-year postoperative failure rate of approximately 40% (PEDIG 2019; Ophthalmology 126: 305-17). For the vast majority of children, surgical failure was due to recurrence of the exodeviation. Only about 30% of treated children had resolution of IXT at the 3-year visit. Similarly, a literature review of 28 surgical studies that included 2530 children with IXT reported a suboptimal surgical outcome at 1-year post-op in approximately 40% of children. (Coffey et al 1992; Optom Vis Sci 69: 386-404).

Poor surgical results for IXT are thought to occur due to poor sensory status (suppression) or inadequate motor alignment. There are few data on the effects of non-surgical interventions designed to improve sensory status of children undergoing surgery for IXT. Although several retrospective case reviews found evidence supporting a benefit of pre-op sensory and motor fusion training on IXT surgical outcomes, there have been no prospective studies or randomized clinical trials. One of the largest retrospective case series (Cooper & Leyman 1977; Am Orthoptic J 27:61-7) compared 216 patients with IXT who had sensory and motor fusion training prior to surgery with 264 who had surgery alone and found a higher rate of good surgical outcomes (52% vs 42%). There are no published data on post-op interventions to improved sensory status.

In this study, engaging movies will be presented on a handheld Nintendo to decrease suppression and engage stereoacuity. In previous research, use of dichoptic games and movies by children with amblyopia has been shown to reduce suppression and encourage sensory fusion (Birch et al 2015, JAAPOS 19:6-11; Birch et al 2019, JAAPOS [Epub ahead of print]; Kelly, Jost, et al 2016; JAMA Ophthalmol 134:1402-8.; Kelly et al Invest 2018 Ophthalmol Vis Sci 59:1221-8; Li et al 2014; Eye 28: 1246-53). This approach will be adapted by using dichoptic movies presented on a Nintendo for children with IXT to improve their stereoacuity and reduce their suppression in an effort improve control of alignment sufficiently without surgery (Aim 1) or to improve stability of post-operative alignment (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IXT
* IXT control assessment score at distance of 3 or 4 at baseline
* Ocular misalignment by PACT >10 pd at distance and near or PACT >15 at distance or near

Exclusion Criteria:

* Amblyopia
* Prior surgery
* Prior binocular treatment
* Coexisting ocular or systemic condition
* Developmental delay

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Alignment Control Score | 3 months
  Classification system developed by PEDIG to quantify the degree of control of ocular alignment on a 0-5 scale at distance and near; 0 is best control [no exotropia unless dissociated, recovers in <1 second (phoria)] and 5 is worst control (constant exotropia)

SECONDARY OUTCOMES:
Stereoacuity at distance | 3 months
  Randot Distance Stereoacuity Test
Binocular fixation stability | 3 months
  Stability of the vergence angle assessed by recording eye movements during 20 sec fixation
Stereoacuity at near | 3 months
  Randot Preschool Stereoacuity Test

CONTACTS AND LOCATIONS:
Overall Officials: Eileen E Birch, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Eileen E Birch, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No